CLINICAL TRIAL: NCT04779450
Title: The Effect of Telemonitoring on Upper Limb Function, Quality of Life and Risk of Lymphedema During and After Pandemic COVID-19 in Women Submitted to Treatment for Breast Cancer: A Randomized Controlled Trial
Brief Title: Effect of Telemonitoring on Functionality, Quality of Life and Risk of Lymphedema in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Gilmar Moraes Santos, PT, Clinical Teacher, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Telemonitoring BCS
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Synchronous Telemonitoring (Experimental): The sessions will be supervised by a therapist and conducted via video call using the WhatsApp® application, lasting 50 minutes, 3 times a week, for 6 consecutive weeks, the exercises will basically consist of active stretching, mobilization and scapular stabilization, and active shoulder exercises with gradual range of motion.
  Interventions: Other: Kinesiotherapy protocol
- Asynchronous Telemonitoring (Experimental): An explicative schedule with the exercises to be performed asynchronously during the week will be delivered weekly via e-mail and WhatsApp®. The exercises will be the same as those performed by the synchronous telemonitoring group, and the participant will be free to ask any questions about the protocol to the therapist at any time via text message or e-mail.
  Interventions: Other: Kinesiotherapy protocol
- Control Group (Active Comparator): Will receive only a booklet of usual guidelines for women after breast cancer, such as skin care, return to activities, upper limb functionality, self-care, lymphedema and physical activity practice.
  Interventions: Other: Usual orientations

INTERVENTIONS:
Other: Kinesiotherapy protocol — The kinesiotherapy protocol is an exercise-based treatment designed to gain upper limb range of motion and muscle strengthening.
  Arms: Asynchronous Telemonitoring; Synchronous Telemonitoring
Other: Usual orientations — Usual orientations for post-breast cancer women, such as skin care, return to activities, upper limb functionality, self-care, lymphedema, and physical activity practice.
  Arms: Control Group

SUMMARY:
The objective of the study is to evaluate the effectiveness of telemonitoring in the dysfunctions of the upper limbs in activities of daily living, quality of life and prevention of lymphedema in women undergoing treatment for breast cancer. Secondarily, to analyze the degree of satisfaction in the proposed treatment modality. This is a randomized controlled trial, double blind (evaluator and patient), parallel in three groups (synchronous telemonitoring group, asynchronous telemonitoring group and control group). The protocol will last six weeks, and quality of life, upper limb functionality, and risk of lymphedema will be evaluated. Both intervention groups will be submitted to a kinesiotherapy program three times a week, with synchronous and asynchronous monitoring, while the control group will receive usual post cancer orientations. Kinesiotherapy protocol in synchronous form compared to the usual recommendations in remote form is expected to show superior result in upper limb function and quality of life of women after breast cancer.

DETAILED DESCRIPTION:
This is a randomized, double blind (evaluator and patient), parallel control trial in three groups (synchronous telemonitoring group, asynchronous telemonitoring group, and control group). The allocation of the participants will be done by an external member, through a masked draw, the name of each participant will be in numbered opaque envelopes, which will only be opened after the initial evaluation, to blind the evaluating therapist, a second therapist will be responsible for the application of the interventions. The protocol for the intervention groups will last 6 weeks, and the exercises will basically consist of active stretching, mobilization and scapular stabilization, and active shoulder exercises with gradual range of motion. The intervention was based on previous studies that used standard kinesiotherapy in their outcomes.

The sessions for the synchronous telemonitoring group will be supervised and conducted via video call using the WhatsApp® application, lasting 50 minutes, 3 times a week.

For the asynchronous telemonitoring group, an explanatory schedule with the exercises to be performed during the week will be delivered weekly via e-mail and WhatsApp®. The exercises will be the same as those performed by the previous group, and the participant will be free to ask any questions about the protocol with the therapist at any time via text message or e-mail. The control group will receive only the usual orientation booklet for post-breast cancer women. The participants who agree to participate in the research will sign the Informed Consent Form, and may withdraw from the research at any stage of the study. Assessment and intervention collection will take place via video call. The personal identification data of the participants will be preserved in accordance with the resolution of the national health council, taking into account the possibility of scientific dissemination of the results obtained. The selection method adopted will be non-probability sampling, convenience sampling. The participants of the study will be recruited in the reference hospital for oncologic care in Florianópolis- State of Santa Catarina/Brazil, the Oncology Research Center, through a retrospective and active search in the medical records, in order to recover clinical data and contact of the participants with up to 24 months after the curative surgical intervention. There will also be recruitment through dissemination of the study via media and social networks, folders and messages, so that women voluntarily apply for the research. The sample will consist of women diagnosed with breast cancer and undergoing surgical treatment, with up to 24 months postoperatively, present functional disability and impaired quality of life, able to understand and access mobile applications or live with someone who helps them, have access to the internet and telephone for contact.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18;
* Diagnosed with breast cancer and submitted to surgical treatment, regardless of the type of surgery;
* With up to 24 months post-operatively, already completed cycles of adjuvant therapies (radiotherapy and/or chemotherapy);
* Moderate functional disability with a minimum score of 30% QuickDash questionnaire;
* Impaired quality of life;
* Able to understand and access mobile applications or live with someone who assists, has internet access and telephone contact.

Exclusion Criteria:

* open lesions;
* acquired infections;
* chronic disease or previous motor sequelae that would interfere with participation in the study;
* women who have difficulty understanding the questions or questionnaires applied or proposed activities;
* diagnosis of lymphedema;
* have no functional alterations in the upper limbs or quality of life.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Upper Limb Functionality | Change in Quick DASH total score Pre-intervention at 6 weeks Post-intervention
  Quick Disabilities of the Arm, Shoulder and Hand (DASH) is an 11-item questionnaire designed to assess the physical disability and symptoms of the upper limbs during activities of daily living, during the week prior to the assessment. The questions are scored from 1 to 5, where 1 corresponds to "no difficulty" and 5 "could not do", and the higher the score, the higher the level of disability. The total score is 100 points, is calculated by adding the first total of answers, then dividing that number by the total number of items answered, this value is subtracted by 1 and multiplied by 25.
Assessment of quality of life | Change in EORTC QLQ BR-23 total score Pre-intervention at 6 weeks Post-intervention
  European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life Questionnaire BR-23 was developed in 1996 by the European Organization for Research and Treatment of Cancer (EORTC) specifically to assess quality of life in patients with breast cancer. The EORTC QLQ-BR-23 comprises 23 questions and assesses the symptoms experienced in the last week, and has two domains (functional and symptoms). The answers are displayed on a Likert scale, with values from 1 to 4, in which case the higher the final score, the better the quality of life.

SECONDARY OUTCOMES:
Arm circumference | Change from Pre Intervention Circumference of the arm at 6 weeks Post Intervention
  The circumference of the arm will be evaluated by the perimeter.
Level of satisfaction | 6 weeks Post Intervention
  Evaluated qualitatively and quantitatively, addressed only at the re-evaluation period questions such as, " How was your experience with this treatment modality?", "From zero to ten, how much would you recommend this treatment modality?", "From zero to ten, how satisfied were you with this intervention?"

CONTACTS AND LOCATIONS:
Overall Officials: Gilmar M Santos, PhD, Study Chair — university of santa catarina state
Locations (1):
- Santa Catarina State University, Florianópolis, Santa Catarina, Brazil